CLINICAL TRIAL: NCT04501913
Title: Remote Perioperative Telemonitoring of Patient-Generated Physiologic Health Data and Patient-Reported Outcomes
Brief Title: Remote Telemonitoring of Patient-Generated Physiologic Health Data and Patient-Reported Outcomes
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19040; NCI-2020-03377 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19040 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-05-21; First posted 2020-08-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Clinical Stage 0 Esophageal Adenocarcinoma AJCC v8; Clinical Stage 0 Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage 0 Gastric Cancer AJCC v8; Clinical Stage I Esophageal Adenocarcinoma AJCC v8; Clinical Stage I Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage I Gastric Cancer AJCC v8; Clinical Stage II Esophageal Adenocarcinoma AJCC v8; Clinical Stage II Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage II Gastric Cancer AJCC v8; Clinical Stage IIA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IIA Gastric Cancer AJCC v8; Clinical Stage IIB Esophageal Adenocarcinoma AJCC v8; Clinical Stage IIB Gastric Cancer AJCC v8; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage IV Esophageal Adenocarcinoma AJCC v8; Clinical Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IVA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IVA Gastric Cancer AJCC v8; Clinical Stage IVB Esophageal Adenocarcinoma AJCC v8; Clinical Stage IVB Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IVB Gastric Cancer AJCC v8; Hepatobiliary Neoplasm; Malignant Digestive System Neoplasm; Malignant Female Reproductive System Neoplasm; Malignant Genitourinary System Neoplasm; Malignant Neoplasm; Pathologic Stage 0 Esophageal Adenocarcinoma AJCC v8; Pathologic Stage 0 Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage 0 Gastric Cancer AJCC v8; Pathologic Stage I Esophageal Adenocarcinoma AJCC v8; Pathologic Stage I Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage I Gastric Cancer AJCC v8; Pathologic Stage IA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IA Gastric Cancer AJCC v8; Pathologic Stage IB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IB Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IB Gastric Cancer AJCC v8; Pathologic Stage IC Esophageal Adenocarcinoma AJCC v8; Pathologic Stage II Esophageal Adenocarcinoma AJCC v8; Pathologic Stage II Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage II Gastric Cancer AJCC v8; Pathologic Stage IIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IIA Gastric Cancer AJCC v8; Pathologic Stage IIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIB Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IIB Gastric Cancer AJCC v8; Pathologic Stage III Esophageal Adenocarcinoma AJCC v8; Pathologic Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage III Gastric Cancer AJCC v8; Pathologic Stage IIIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IIIA Gastric Cancer AJCC v8; Pathologic Stage IIIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIB Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IIIB Gastric Cancer AJCC v8; Pathologic Stage IIIC Gastric Cancer AJCC v8; Pathologic Stage IV Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IV Gastric Cancer AJCC v8; Pathologic Stage IVA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IVB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IVB Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage I Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage I Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage II Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage II Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage III Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIA Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIA Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIB Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIB Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Esophageal Squamous Cell Carcinoma AJCC v8; Stage 0 Colorectal Cancer AJCC v8; Stage 0a Bladder Cancer AJCC v8; Stage 0is Bladder Cancer AJCC v8; Stage I Bladder Cancer AJCC v8; Stage I Cervical Cancer AJCC v8; Stage I Colorectal Cancer AJCC v8; Stage I Ovarian Cancer AJCC v8; Stage I Prostate Cancer AJCC v8; Stage I Renal Cell Cancer AJCC v8; Stage I Uterine Corpus Cancer AJCC v8; Stage IA Cervical Cancer AJCC v8; Stage IA Ovarian Cancer AJCC v8; Stage IA Uterine Corpus Cancer AJCC v8; Stage IA1 Cervical Cancer AJCC v8; Stage IA2 Cervical Cancer AJCC v8; Stage IB Cervical Cancer AJCC v8; Stage IB Ovarian Cancer AJCC v8; Stage IB Uterine Corpus Cancer AJCC v8; Stage IB1 Cervical Cancer AJCC v8; Stage IB2 Cervical Cancer AJCC v8; Stage IC Ovarian Cancer AJCC v8; Stage II Bladder Cancer AJCC v8; Stage II Cervical Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage II Ovarian Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage II Renal Cell Cancer AJCC v8; Stage II Uterine Corpus Cancer AJCC v8; Stage IIA Cervical Cancer AJCC v8; Stage IIA Colorectal Cancer AJCC v8; Stage IIA Ovarian Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIA1 Cervical Cancer AJCC v8; Stage IIA2 Cervical Cancer AJCC v8; Stage IIB Cervical Cancer AJCC v8; Stage IIB Colorectal Cancer AJCC v8; Stage IIB Ovarian Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Colorectal Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage III Bladder Cancer AJCC v8; Stage III Cervical Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage III Renal Cell Cancer AJCC v8; Stage III Uterine Corpus Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8; Stage IIIA Cervical Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIA Uterine Corpus Cancer AJCC v8; Stage IIIA1 Ovarian Cancer AJCC v8; Stage IIIA2 Ovarian Cancer AJCC v8; Stage IIIB Bladder Cancer AJCC v8; Stage IIIB Cervical Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIB Uterine Corpus Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IIIC Uterine Corpus Cancer AJCC v8; Stage IIIC1 Uterine Corpus Cancer AJCC v8; Stage IIIC2 Uterine Corpus Cancer AJCC v8; Stage IV Bladder Cancer AJCC v8; Stage IV Cervical Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Stage IV Uterine Corpus Cancer AJCC v8; Stage IVA Bladder Cancer AJCC v8; Stage IVA Cervical Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVA Uterine Corpus Cancer AJCC v8; Stage IVB Bladder Cancer AJCC v8; Stage IVB Cervical Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8; Stage IVB Uterine Corpus Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Gastrointestinal Neoplasms; Urogenital Neoplasms; Neoplasms; Colorectal Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Carcinoma, Renal Cell | interventions — Remote Patient Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (remote telemonitoring): Patients undergo remote perioperative telemonitoring with home monitoring devices activity monitor beginning 7 days before surgery and up to 30 days after hospital discharge.
  Interventions: Procedure: Patient Monitoring; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Patient Monitoring — Undergo remote perioperative telemonitoring
  Other Names: medical monitoring; monitor
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study examines at-home monitoring of patient-generated phsyiologic health data and patient-reported outcomes. Patient-generated health data using at-home monitoring devices and smart device applications are used more and more to measure value and quality in cancer care. This trial may show whether at-home monitoring programs can improve the care of patients after hospital discharge from surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility and acceptability of remote perioperative monitoring in solid tumor cancer patients scheduled for gastrointestinal (GI), genitourinary (GU), gynecological (GYN) cancer surgery.

II. To explore patterns, trajectory, and changes in physiologic health parameter outcomes (weight, temperature, oxygen saturation, heart rate, blood pressure, daily steps) and patient-reported outcomes (PROs) (symptoms, quality of life [QOL]) from pre-surgery to the post-discharge period.

III. To explore the relationship between changes in physiologic health parameter outcomes/PROs and surgical outcomes (postoperative complications, readmissions).

IV. To explore changes in physiologic health parameters and PROs by open surgery versus minimally invasive (laparoscopic or robotic) surgery.

OUTLINE:

Patients undergo remote perioperative telemonitoring with home monitoring devices activity monitor beginning 7 days before surgery and up to 30 days after hospital discharge.

After completion of study, patients are followed up for 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients diagnosed with GI (esophagus, gastric, colorectal, hepatobiliary) GU (prostate, bladder, renal cell), or GYN (ovarian, endometrial, cervical) cancers
* Patients who are scheduled to undergo major abdominal/pelvic surgery for cancer treatment
* Ability to read and understand English
* We are targeting patients across all stages of disease
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients diagnosed with gastrointestinal, genitourinary, or gynecological cancers who are scheduled to undergo abdominal/pelvic surgery at the City of Hope National Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Overall accrual | Days 2
  Planned accrual is bound by the number of eligibile patients and duration of the study funding. Accrual goal is 20 patients.
Overall accrual | Days 7
  Planned accrual is bound by the number of eligibile patients and duration of the study funding. Accrual goal is 20 patients.
Overall accrual | Days 14
  Planned accrual is bound by the number of eligibile patients and duration of the study funding. Accrual goal is 20 patients.
Overall accrual | Days 30 after discharge
  Planned accrual is bound by the number of eligibile patients and duration of the study funding. Accrual goal is 20 patients.
Retention | Days 2
  Participants' retention will be assessed at all follow-up timepoints by remaining enrolled on study.
Retention | Days 7
  Participants' retention will be assessed at all follow-up timepoints by remaining enrolled on study.
Retention | Days 14
  Participants' retention will be assessed at all follow-up timepoints by remaining enrolled on study.
Retention | Days 30 after discharge
  Participants' retention will be assessed at all follow-up timepoints by remaining enrolled on study.
Attrition rates | Days 2
  All participants that are enrolled will be tracked and assessed for drop off (attrition) at all time points.
Attrition rates | Days 7
  All participants that are enrolled will be tracked and assessed for drop off (attrition) at all time points.
Attrition rates | Days 14
  All participants that are enrolled will be tracked and assessed for drop off (attrition) at all time points.
Attrition rates | Days 30 after discharge
  All participants that are enrolled will be tracked and assessed for drop off (attrition) at all time points.
Patient's ability to use the remote perioperative monitoring equipment | Up to 30 days
  At least 75% of patients will be able to wear the wristband pedometer for at least 1 week post-operatively, and at least 75% of the patients will be able to use at least 2 out of 4 physiologic devices (scale, pulse/heart monitor, blood pressure cuff, and thermometer) at least once a week.
Staff ability to identify threshold healthcare parameters | Up to 30 days
  Staff will be alerted through a workflow guided by the threshold healthcare parameters. The number of alerts of data outside parameters will be recorded as well as the initiated response to each alert.
Staff ability to act on identified threshold healthcare parameters | Up to 30 days
  The number of alerts and resolved alerts will be captured in response to threshold parameters in addition to a nurse debriefing form to summarize the response

SECONDARY OUTCOMES:
Patterns, trajectory, and changes in patient-generated health data (PGHD) | Up to 30 days
  After discharge, all patient-generated physiologic data will be repeated at day 7,14,,and day 30 to measure any differences in weight, temperature, oxygen saturation, heart rate, blood pressure and functional activity using the Aetonix devices and Vivofit watches
Patient reported outcomes (PROs) (symptoms, quality of life [QOL]) between groups | From pre-surgery to the post-discharge period
  Quality of Life will be measured through the EQ-5D-5L and PROMIS 4 QOL measurement tools
Changes in PGHD/PROs | Up to 30 days after surgery
  Distributions of PGHD/PROs will be generated. Means, standard deviations, and ranges will be calculated for continuous variables, and frequencies and percentages for categorical variables. All PROs will be scored according to instructions. Analysis of variance (ANOVA) will be used to study patterns of change over time in PROs administered at multiple time points.

CONTACTS AND LOCATIONS:
Overall Officials: Laleh Melstrom, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States